CLINICAL TRIAL: NCT05913622
Title: Randomized Embedded Multifactorial Adaptive Platform in ExtraCorporeal Membrane Oxygenation (REMAP ECMO) - Left Ventricular Unloading Study
Brief Title: A Study on the Effects of Left Ventricular Unloading in the Setting of VA ECMO Support
Acronym: REMAP ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, Christiaan Meuwese, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82979.078.23
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cardiogenic Shock
Keywords: Left ventricular unloading; Venoarterial ExtraCorporeal Membrane Oxygenation (VA ECMO); Cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Intervention Model Description: Adaptive Bayesian Platform Trial evaluating multiple interventions in multiple domains
Masking Description: No masking is possible as the device is visible after placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IABP unloading arm (Experimental): This group of patients will receive an intra-aortic balloon pump (IABP) as an adjunct to VA ECMO support. When allocated to the IABP unloading arm, patients must receive an IABP within 8 hours after VA ECMO initiation.
  Interventions: Device: Intra-aortic balloon pump
- ECMO alone arm (No Intervention): This group of patients will receive VA ECMO support without left ventricular unloading device after randomization.

INTERVENTIONS:
Device: Intra-aortic balloon pump — An IABP is placed percutaneously into the thoracic aorta and supports the heart through synchronized inflation and deflation of a balloon.
  Other Names: IABP
  Arms: IABP unloading arm

SUMMARY:
REMAP ECMO is a registry based platform in which multiple response adaptive randomized clinical trials (trial domains) will be embedded. These trial domains will, in a perpetual way, study the effects of a range of patient management strategies which aim to improve VA ECMO weaning success. A first trial domain will address the effects of left ventricular (LV) unloading through intra-aortic balloon pumping on weaning succes in VA ECMO supported patients.

DETAILED DESCRIPTION:
ExtraCorporeal Membrane Oxygenation (ECMO) is increasingly used but remains associated with high weaning failure- and mortality- rates. This seems in part attributable to a knowledge gap on how to properly manage ECMO and its related therapies as current knowledge and treatment protocols are based on observational studies and expert opinions. The "Randomized Embedded Multifactorial Adaptive Platform in ECMO" (REMAP ECMO) study was developed to study, in an efficient and randomized way, different ECMO related patient management issues and will consist of two parts:

1. A patient registry that will serve for quality monitoring and observational studies of ECMO patients being treated in participating centers.
2. Embedded within the registry, multiple response adaptive randomized clinical trials (trial domains) which aim to evaluate the effectiveness of a range of therapeutic interventions on ECMO weaning success. These interventions all have in common that they are all already used in ECMO care but their use depends on center and/or doctors preferences as no high quality (randomized) evidence guiding their indication, timing and management exists.

   * LV unloading trial A first trial domain to be initiated within the REMAP ECMO platform will address the effects of left ventricular (LV) unloading, through application of an intra-aortic balloon pump (IABP), on weaning success in the setting of venoarterial (VA) ECMO. The rationale of this trial domain is based on the increase in LV loading conditions, as induced by VA ECMO, which could lead to pulmonary edema, intracardiac thrombosis and even death. These serious sequelae could possibly be prevented by adding IABP as adjunct to VA ECMO therapy.
   * Physiological substudy on IABP as adjunct to V-A ECMO

A nested physiological observational substudy within the ongoing REMAP ECMO RCT, using the trial arms where patients are randomized between receiving V-A ECMO with or without IABP in the Erasmus Medical Center Rotterdam. The substudy aims to evaluate the physiological effects of IABP in conjunction with V-A ECMO on respiratory and hemodynamic parameters. The substudy consists of two parts:

1. Microcirculation and Macrocirculation: This part investigates the impact of IABP on both microcirculation and macrocirculation in the setting of V-A ECMO.
2. PEEP as an Unloading Modality: This part examines the effect of Positive End-Expiratory Pressure (PEEP) as an unloading modality during a decremental PEEP trial in patients receiving V-A ECMO, either with or without IABP.

Endpoints in both substudies that can be assessed blindly will be evaluated by an assessor who is blinded to the assigned treatment arm and the objectives of the substudy

ELIGIBILITY:
Inclusion criteria for the registry backbone:

* Having received ECMO support for severe circulatory and/or respiratory insufficiency

Inclusion Criteria for the LV unloading trial domain (VA ECMO + IABP vs VA ECMO alone):

* Cardiogenic shock
* Having received VA ECMO support for severe circulatory (and respiratory insufficiency).
* Age ≥ 18 years
* Initiation of LV unloading (IABP or Impella) possible ≤ 8 hours after ECMO initiation

Exclusion criteria for the registry backbone

* Objection to participation in the registry by the patient and/or proxy
* VA ECMO usage confined to the period during surgery or another intervention (the VA ECMO was removed at the end of the intervention in the operation room).

Exclusion criteria for the LV unloading trial domain (VA ECMO + IABP vs VA ECMO alone)

* No (deferred) informed consent provided by the patient and/or proxy.
* Pregnancy
* ECMO usage confined to the period during surgery or another intervention (the ECMO was removed at the end of the intervention).
* Isolated right ventricular failure (e.g. due to pulmonary embolism).
* Left ventricular assist device (LVAD), Impella or IABP in situ.
* Ventricular septal defect or papillary muscle rupture as the cause of shock.
* Thoracic or abdominal aortic dissection.
* Moderate or severe aortic regurgitation
* Mechanical prosthesis in mitral valve position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
ECMO weaning success | 30 days
  Proportion of patients successfully weaned from VA ECMO at 30 days being defined by; a) being alive, b) without ECMO, IABP or Impella support, and c) not having received a heart transplantation or left ventricular assist device (LVAD).
Physiological substudy: End diastolic volume | within 24 hours after ECMO initiation
  End diastolic volume as assessed by echocardiography

SECONDARY OUTCOMES:
Treatment failure | During ECMO support
  The proportion of patients in whom LV unloading therapy was escalated. Escalation is defined by the insertion of an IABP (only in the VA ECMO alone arm), or Impella or left vent (IABP unloading arm or VA ECMO alone arm).
30 day, 90 day and 1 year mortality | 30 days, 90 days and 1 year after ECMO initiation
  Mortality rate at 30 days, 90 days and 1 year after ECMO initiation
ECMO support duration | Until 30 days after ECMO initiation
  The duration of ECMO support in days
Major bleeding events | Until 30 days after ECMO initiation
  The occurrence of major bleeding events (fatal, in a critical area (intracranial, intraspinal, or intraocular), requiring intervention (coiling or surgery) and/or transfusion of ≥3 packed cells) until 30 days after VA ECMO initiation.
Unplanned surgical or catheter based intervention of the leg(s) | Until 30 days after ECMO initiation
  Unplanned surgical or catheter based intervention of the leg(s) in which ECMO and/or IABP or Impella was inserted until 30 days after ECMO initiation.
Time to lactate normalization | Until 30 days after ECMO initiation
  Time to lactate normalization (<2 mmol/L).
Time to first negative net fluid balance | Until 30 days after ECMO initiation
  Time to first negative net fluid balance (calculated per 24 hours).
The occurrence of continuous venovenous hemofiltration initiation during ECMO support | Until 30 days after ECMO initiation
  The occurrence of continuous venovenous hemofiltration (dialysis) (CVVH(D)) initiation during ECMO support.
Course in PF ratio | Until 30 days after ECMO initiation.
  Course in PaO2/FiO2 (PF) ratio (PaO2 divided by FiO2 provided)
Duration of mechanical ventilation. | Until 30 days after ECMO initiation.
  Duration of mechanical ventilation. Patients on mechanical ventilation via tracheostomy need to be 24 hours free of mechanical ventilation.
Left ventricular ejection fraction 30 days after ECMO initiation. | At 30 days after ECMO initiation.
  Left ventricular ejection fraction 30 days after ECMO initiation.
Time course in vasoactive inotropic score (VIS) during ECMO support | Until 30 days after ECMO initiation.
  Time course in vasoactive inotropic score (VIS) during ECMO support
Time course in NT-pro BNP during ECMO support. | Until 30 days after ECMO initiation.
  Time course in NT-pro BNP during ECMO support.
Quality of life at 1 year | 1 year after ECMO initiation
  Quality of life on basis of EQ5D questionnaires
Total health care costs | 6 and 12 months after ECMO initiation
  Total healthcare costs in euros are determined by using the International Medical Consumption Questionnaire (iMCQ) and the calculated costs after 6 and 12 months of follow up
Hospital readmission rate | 1 year
  The number of hospital readmissions based on the information provided in the international Medical Consumption Questionnaire (iMCQ)
Physiological substudy: Heart rate | 24 and 48 hours after ECMO initiation
  The average heart rate measured during 5 minutes
Physiological substudy: pulmonary artery catheter parameters | 24 and 48 hours after ECMO initiation
  pulmonary artery catheter parameters: pulmonary capillary wedge pressure, cardiac output, central venous pressure
Physiological substudy: Echocardiography | 24 and 48 hours after ECMO initiation
  Echocardiography: LV ejection fraction, TAPSE, VTI LVOT
Physiological substudy: microcirculation measurements | 24 and 48 hours after ECMO initiation
  Microcirculation measurements: Perfused vessel density (PVD [mm/mm2], Total vessel density (TVD [mm/mm2]
Physiological substudy: respiratory parameters | 24 and 48 hours after ECMO initiation
  Respiratory: FiO2, PEEP, Respiratory System Compliance (CRS) as the ratio between Vt/Dp.
Physiological substudy: delta NT-pro BNP | 24 and 48 hours after ECMO initiation
  delta NT-pro BNP

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Meuwese, Principal Investigator — Erasmus Medical Center
Locations (14):
- Belgium (3):
  - AZ Sint-Jan Brugge, Bruges
  - ZOL Genk, Genk
  - UZ Gent, Ghent
- Netherlands (11):
  - Amphia hospital, Breda, North Brabant
  - Catharina hospital, Eindhoven, North Brabant
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haga ziekenhuis, The Hague, South Holland
  - Antonius hospital, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht, Utrecht
  - OLVG, Amsterdam
  - Maastricht UMC, Maastricht
  - Radboud UMC, Nijmegen

REFERENCES:
- [Background] Cheng R, Hachamovitch R, Kittleson M, Patel J, Arabia F, Moriguchi J, Esmailian F, Azarbal B. Complications of extracorporeal membrane oxygenation for treatment of cardiogenic shock and cardiac arrest: a meta-analysis of 1,866 adult patients. Ann Thorac Surg. 2014 Feb;97(2):610-6. doi: 10.1016/j.athoracsur.2013.09.008. Epub 2013 Nov 8. PMID 24210621
- [Background] Keebler ME, Haddad EV, Choi CW, McGrane S, Zalawadiya S, Schlendorf KH, Brinkley DM, Danter MR, Wigger M, Menachem JN, Shah A, Lindenfeld J. Venoarterial Extracorporeal Membrane Oxygenation in Cardiogenic Shock. JACC Heart Fail. 2018 Jun;6(6):503-516. doi: 10.1016/j.jchf.2017.11.017. Epub 2018 Apr 11. PMID 29655828
- [Background] Schrage B, Becher PM, Bernhardt A, Bezerra H, Blankenberg S, Brunner S, Colson P, Cudemus Deseda G, Dabboura S, Eckner D, Eden M, Eitel I, Frank D, Frey N, Funamoto M, Gossling A, Graf T, Hagl C, Kirchhof P, Kupka D, Landmesser U, Lipinski J, Lopes M, Majunke N, Maniuc O, McGrath D, Mobius-Winkler S, Morrow DA, Mourad M, Noel C, Nordbeck P, Orban M, Pappalardo F, Patel SM, Pauschinger M, Pazzanese V, Reichenspurner H, Sandri M, Schulze PC, H G Schwinger R, Sinning JM, Aksoy A, Skurk C, Szczanowicz L, Thiele H, Tietz F, Varshney A, Wechsler L, Westermann D. Left Ventricular Unloading Is Associated With Lower Mortality in Patients With Cardiogenic Shock Treated With Venoarterial Extracorporeal Membrane Oxygenation: Results From an International, Multicenter Cohort Study. Circulation. 2020 Dec;142(22):2095-2106. doi: 10.1161/CIRCULATIONAHA.120.048792. Epub 2020 Oct 9. PMID 33032450
- [Background] Thiele H, Zeymer U, Thelemann N, Neumann FJ, Hausleiter J, Abdel-Wahab M, Meyer-Saraei R, Fuernau G, Eitel I, Hambrecht R, Bohm M, Werdan K, Felix SB, Hennersdorf M, Schneider S, Ouarrak T, Desch S, de Waha-Thiele S; IABP-SHOCK II Trial (Intraaortic Balloon Pump in Cardiogenic Shock II) Investigators; IABP-SHOCK II Investigators. Intraaortic Balloon Pump in Cardiogenic Shock Complicating Acute Myocardial Infarction: Long-Term 6-Year Outcome of the Randomized IABP-SHOCK II Trial. Circulation. 2019 Jan 15;139(3):395-403. doi: 10.1161/CIRCULATIONAHA.118.038201. Epub 2018 Nov 11. PMID 30586721
- [Background] Grandin EW, Nunez JI, Willar B, Kennedy K, Rycus P, Tonna JE, Kapur NK, Shaefi S, Garan AR. Mechanical Left Ventricular Unloading in Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation. J Am Coll Cardiol. 2022 Apr 5;79(13):1239-1250. doi: 10.1016/j.jacc.2022.01.032. PMID 35361346
- [Background] Russo JJ, Aleksova N, Pitcher I, Couture E, Parlow S, Faraz M, Visintini S, Simard T, Di Santo P, Mathew R, So DY, Takeda K, Garan AR, Karmpaliotis D, Takayama H, Kirtane AJ, Hibbert B. Left Ventricular Unloading During Extracorporeal Membrane Oxygenation in Patients With Cardiogenic Shock. J Am Coll Cardiol. 2019 Feb 19;73(6):654-662. doi: 10.1016/j.jacc.2018.10.085. PMID 30765031
- [Background] Na SJ, Yang JH, Yang JH, Sung K, Choi JO, Hahn JY, Jeon ES, Cho YH. Left heart decompression at venoarterial extracorporeal membrane oxygenation initiation in cardiogenic shock: prophylactic versus therapeutic strategy. J Thorac Dis. 2019 Sep;11(9):3746-3756. doi: 10.21037/jtd.2019.09.35. PMID 31656647
- [Derived] van Steenwijk MPJ, van Rosmalen J, Elzo Kraemer CV, Donker DW, Hermens JAJM, Kraaijeveld AO, Maas JJ, Akin S, Montenij LJ, Vlaar APJ, van den Bergh WM, Oude Lansink-Hartgring A, de Metz J, Voesten N, Boersma E, Scholten E, Beishuizen A, Lexis CPH, Peperstraete H, Schiettekatte S, Lorusso R, Gommers DAMPJ, Tibboel D, de Boer RA, Van Mieghem NMDA, Meuwese CL; REMAP ECMO LV unloading study group. A randomized embedded multifactorial adaptive platform for extra corporeal membrane oxygenation (REMAP ECMO) - design and rationale of the left ventricular unloading trial domain. Am Heart J. 2025 Jan;279:81-93. doi: 10.1016/j.ahj.2024.10.010. Epub 2024 Oct 22. PMID 39447716